CLINICAL TRIAL: NCT06059911
Title: The Effect of a Pre-workout Supplement on Basketball-specific Performance and Biochemical Profile of Well-trained Athletes
Brief Title: Pre-workout Supplementation and Basketball
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Athanasios Z. Jamurtas (Other)
Responsible Party: Sponsor-Investigator, Athanasios Z. Jamurtas, Professor, University of Thessaly
Organization: University of Thessaly (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Douligeris Study
Record Dates: First submitted 2023-09-15; First posted 2023-09-29 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Sport Performance
MeSH Terms: interventions — Caffeine; Creatine; citrulline malate; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multi-ingredient dietary supplement (Experimental): 20 g of a multi-ingredient dietary supplement. Composition: 200 mg caffeine, 3.3 g creatine monohydrate, 3.2 g β-alanine, 6 g citrulline malate and 5 g BCAA
  Interventions: Dietary Supplement: Multi-ingredient dietary supplement (caffeine, creatine monohydrate, β-alanine, citrulline malate, BCAA)
- Placebo dietary supplement (97% maltodextrin) (Placebo Comparator): 20 g of isoenergetic placebo dietary supplement. Composition: 97% flavored maltodextrin, similar in color, flavor, taste and energy to the experimental multi-ingredient supplement
  Interventions: Dietary Supplement: Placebo dietary supplement (97% maltodextrin)

INTERVENTIONS:
Dietary Supplement: Multi-ingredient dietary supplement (caffeine, creatine monohydrate, β-alanine, citrulline malate, BCAA) — Administration of a multi-ingredient dietary supplement consisting of 200 mg caffeine, 3.3 g creatine monohydrate, 3.2 g β-alanine, 6 g citrulline malate and 5 g branched chain amino acids
  Arms: Multi-ingredient dietary supplement
Dietary Supplement: Placebo dietary supplement (97% maltodextrin) — Administration of an isoenergetic placebo comparator dietary supplement consisting of 97% maltodextrin
  Arms: Placebo dietary supplement (97% maltodextrin)

SUMMARY:
Pre-workout supplements (PWS) consumption in recreationally or physically trained males lead to many performance-enhancing benefits, including improvements in mean power output during single and repeated sprints, agility, reaction times, lower body muscular endurance and reduced fatigue. PWS ingestion also improves anaerobic performance and prolongs time to exhaustion during high-intensity intermittent exercise. However, PWSs' effectiveness is not constant, as they do not alter anaerobic power, jumping performance or blood lactate concentrations after a training session, at least in recreationally trained males and strength-power athletes. Moreover, the effects of long-term PWS supplementation, where some nutritional agents were combined (e.g., β-alanine, creatine, citrulline malate, etc.) to assess endurance-trained runners or elite cyclists' performance, are mixed and less clear. Even though the popularity of PWS use has increased among trained/professional athletes, most of the data in this area are derived from recreationally and not from well-trained athletes of a competitive level (especially in team sports). Therefore, the present study aimed to examine the acute and chronic effects of a PWS, containing 200 mg caffeine, 3.3 g creatine monohydrate, 3.2 g βalanine, 6 g citrulline malate and 5 g BCAA per dose, on shooting, jumping, sprinting, agility, aerobic and anaerobic performance in well-trained basketball players.

DETAILED DESCRIPTION:
According to a randomized, double-blind, placebo-controlled, research design, 36 well-trained male basketball players will be recruited. During their first visit, they will complete a health history and exercise questionnaire and will sign a written informed consent. Participants' dietary profile will be evaluated using 3- day diet recalls and they will be instructed to follow the same dietary scheme for 3 days prior to the subsequent evaluations. During the second visit, participants will be familiarized with the performance evaluations (shooting, jumping, sprinting, agility, running-based anaerobic sprint test and Yo-Yo intermittent recovery level 1 test).

(Acute phase) One week later, Moreover, they will randomly be assigned in two groups (PWS and placebo) by a research member not involved in data collection. After that participants will visit the basketball court in the morning and a blood sample will be collected after overnight fasting. Afterward, the participants in each group will perform the evaluations without PWS or PL. The evaluations will be performed according to National Strength and Conditioning Association standards. Body composition, resting heart rate, blood pressure, basketball-specific shooting exercise, counter-movement jump, 20-m sprint, agility T-Test, running-based anaerobic sprint test and Yo-Yo intermittent recovery level 1 test. One week later, all participants will visit the same basketball court at the same hour and will consume the PWS or placebo supplement and 30 minutes later their physiological characteristics and performance will be evaluated in the same sequence.

(Chronic phase) Following the evaluations of the acute phase, participants will continue the consumption of the PWS or placebo, according to their allocation group, daily for a period of 4 weeks. At the end of the supplementation period, participants will visit the basketball court and a second blood sample will be collected after overnight fasting (the first blood sample, collected before the acute phase evaluations, will serve as baseline). Then, participants' performance will be evaluated in the same sequence as the previous visit.

ELIGIBILITY:
Inclusion Criteria:

1. Male participants, 18-41 years old
2. Absence of drugs, abuse or medications, which are known to affect the Shooting, sprinting, jumping, agility, anaerobic and endurance performance
3. Consent to follow a regular dietary plan for basketball players

Exclusion Criteria:

1. Restraining orthopedic/neuromuscular problems
2. Caffeine hypersensitivity
3. Consumption of more than three servings of coffee per day
4. Use of any supplement or steroids prior to the study
5. Use of creatine, β-alanine, citrulline malate or BCAA-protein supplementation at least six months before the initiation of the study

Ages: 18 Years to 41 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-12-15 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
Countermovement jump height | baseline and up to 4 weeks
  Jumping performance will be evaluated using a contact platform
20 meters sprint running time | baseline and up to 4 weeks
  Sprint performance will be evaluated using photocell gates
Rate of agility T-test performance | baseline and up to 4 weeks
  Agility T-test will be evaluated using photocell gates
Rate of running-based anaerobic sprint test performance | baseline and up to 4 weeks
  Running-based anaerobic sprint test performance will be evaluated using photocell gates
Rate of Yo-Yo intermittent recovery test level 1 test performance | baseline and up to 4 weeks
  Yo-Yo intermittent recovery test level 1 test performance will be evaluated using a field-based test
Rate of basketball-specific shooting performance | baseline and up to 4 weeks
  Basketball-specific shooting performance will be evaluated with a test consisting of 30 free shoots, 30 middle-distance shoots and 30 long-distance shoots
Blood lactate concentartion | baseline and up to 4 weeks
  Blood lactate concentration will be measured using a portable blood lactate analyzer
Creatine kinase concentration | baseline and up to 4 weeks
  Creatine kinase activity will be measured on a clinical chemistry analyzer
Lactate dehydrogenase concentration | baseline and up to 4 weeks
  Lactate dehydrogenase will be measured on a clinical chemistry analyzer
Alkaline phosphatase concentration | baseline and up to 4 weeks
  Alkaline phosphatase will be measured on a clinical chemistry analyzer
Gamma-glutamyltransferase concentration | baseline and up to 4 weeks
  Gamma-glutamyltransferase will be measured on a clinical chemistry analyzer
Urea concentration | baseline and up to 4 weeks
  Urea will be measured on a clinical chemistry analyzer
Creatinine concentration | baseline and up to 4 weeks
  Creatinine will be measured on a clinical chemistry analyzer
Serum glutamic-oxaloacetic transaminase activity | baseline and up to 4 weeks
  Serum glutamic-oxaloacetic transaminase will be measured on a clinical chemistry analyzer
Serum glutamate-pyruvate transaminase activity | baseline and up to 4 weeks
  Serum glutamate-pyruvate transaminase will be measured on a clinical chemistry analyzer

SECONDARY OUTCOMES:
Body mass | baseline and up to 4 weeks
  Body mass will be measured using a calibrated digital scale
Body height | baseline and up to 4 weeks
  Body height will be measured using a stadiometer
Body fat mass | baseline and up to 4 weeks
  Body fat mass will be measured using a calibrated digital scale via bioelectrical impedance analysis
Systolic and diastolic blood pressure | baseline and up to 4 weeks
  Systolic and diastolic blood pressure will be measured using a blood pressure monitor
Heart rate | baseline and up to 4 weeks
  Heart rate will be measured using a heart rate monitor

CONTACTS AND LOCATIONS:
Overall Officials: Sousana K Papadopoulou, Study Director — International Hellenic University
Locations (1):
- Sports Nutrition Laboratory, International Hellenic University, Thessaloniki, Greece